CLINICAL TRIAL: NCT01336335
Title: The Effects of Continuous Positive Airway Pressure (CPAP) on Sympathetic Activity in Different Sites of Activation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Geraldo Lorenzi-Filho, Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sympathetic activity and OSA
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2010-07

CONDITIONS: Radionuclide Imaging (MIBG Scintigraphy); Exercise Test; Blood Pressure Monitoring, Ambulatory; Sympathetic Nerve Activity; Catecholamines
Keywords: sleep apnea, obstructive; sympathetic nerve activity; treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): OSA treatment with CPAP
  Interventions: Device: CPAP
- control (No Intervention): no intervention

INTERVENTIONS:
Device: CPAP — CPAP
  Arms: CPAP

SUMMARY:
Recent evidences suggest that obstructive sleep apnea (OSA) can contribute to cardiovascular disease even in the absence of hypertension. However, there are few data regarding the impact of OSA on the sympathetic system in apparently normotensive patients with OSA as well as the impact of treatment with continuous positive airway pressure in different sites of activation (heart, peripheral nerves and circulating catecholamines)

ELIGIBILITY:
Inclusion Criteria:

* Severe OSA males

Exclusion Criteria:

* Smoking

  * Sustained Hypertension
  * Heart failure
  * Diabetes
  * Renal diseases
  * Under use of any medication
  * Under treatment for OSA

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
improvement in sympathetic activity in muscle sympathetic nerve activity (MSNA) | 3 months
  Improvement in MSNA will be quantified as burst frequency over time (bursts per minute) and as burst frequency corrected for heart rate values (bursts per 100 heartbeats)in the begining and after 3 months.

SECONDARY OUTCOMES:
improvement in sympathetic activity evaluated in different sites of activation | 3 months
  All measurement will be performed at the begining and after 3 months. Blood: blood and 24 hour urine will be collected for norepinephrine quantification.
  Heart: Early (15 min) and delayed (3 hr) planar images will be taken after injection of (123)I-MIBG. The mean counts of the whole heart and the mediastinum will be obtained to calculate heart-to-mediastinum count ratios from the early images (H/Me) and from the delayed images (H/Md) and the myocardial washout rate (WR).
  Blood pressure: 24 hour ambulatory blood pressure monitoring and blood pressure during exercise test (treadmill test)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Pedrosa, MD, PhD, Principal Investigator — Heart Institute (InCor)
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil